CLINICAL TRIAL: NCT01952496
Title: Load Experienced While Using a Stander in Children With Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gillette Children's Specialty Healthcare (Other)
Collaborators: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15994; 1308M40341 (Other: University of MN Insitutional Review Board)
Record Dates: First submitted 2013-09-17; First posted 2013-09-30 (Estimated); Last update posted 2016-02-17 (Estimated); Status verified 2016-02

CONDITIONS: Cerebral Palsy
Keywords: Cerebral Palsy; Non ambulatory; Neuromuscular disability; Children
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Force-measuring platform (Other): A force-measure platform will be placed under each foot of the subject to record the time course of load borne by each of the lower extremities during weight-bearing training in an assisted standing device.
  Intervention: Assisted Standing Treatment Program. Assisted standing treatment program will include at least 2 hours a day, 5 days a week (a total of at least 10 hours a week) for a period of ~9 months.
  Interventions: Other: Assisted Standing Treatment Program

INTERVENTIONS:
Other: Assisted Standing Treatment Program — Assisted standing treatment program will include at least 2 hours a day, 5 days a week (a total of at least 10 hours a week) for a period of ~9 months.
  Arm: Force-measuring platform

SUMMARY:
The goal of this project is to design and validate a force-measuring platform that will measure the magnitude and duration of the load experienced by the lower extremities of individuals with a neuromuscular disability who use a stationary assisted standing device to increase their Bone Mineral Density.

DETAILED DESCRIPTION:
Non-ambulatory children with a neuromuscular disability are at significant risk for poor bone health as reflected by low bone mineral density (BMD) and increased propensity to fracture. In large part, this is due to abnormally low levels of load experienced by the skeleton. A common approach for increasing BMD is to stimulate the musculoskeletal system by increasing the amount and duration of weight-bearing in the lower extremities. For non-ambulatory individuals, this typically takes the form of using an assisted standing device to enable the child to spend time in a standing position so that their lower limbs can experience some degree of body weight. Some of these physical interventions result in varying degrees of improvement in BMD, and some do not. This lack of clarity in outcomes may result from a failure to objectively measure the magnitude and duration of the load experienced by the lower extremities. A lack of change in BMD may be due to the extremities experiencing only a fraction of the body weight due to load-sharing with the assistive device, or to an inadequate duration of standing time. The goal of this project will be to design and validate a force-measuring platform that will measure the magnitude and duration of the load experienced by the lower extremities of individuals with a neuromuscular disability who use a stationary assisted standing device to increase their BMD.

ELIGIBILITY:
Inclusion Criteria:

1. < 18 years old
2. Diagnosed with Cerebral Palsy (CP)
3. Treated at Gillette Children's Specialty Healthcare
4. Gross Motor Function Classification System level of IV or V (non-ambulatory without assistance)
5. Participating in a standing program using a stationary assisted standing device
6. Parent/Guardian willing and able to give consent

Exclusion Criteria:

None

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 3 (Actual)
Dates: Start 2014-02; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Bone Mineral Density | 12 months
  Bone Mineral Density will be measured via dual energy x-ray absorptiometry (DXA) and peripheral quantitative computed tomography (pQCT) scans.

SECONDARY OUTCOMES:
Weight (load)experienced by lower extremities | 12 months
  A platform will measure the magnitude of the load experienced by the lower extremities of individuals with a neuromuscular disability who use a stationary assisted standing device to increase their Bone Mineral Density.
Duration of standing treatment session(s) (time) | 12 months
  A platform will measure the duration of the load experienced by the lower extremities of individuals with a neuromuscular disability who use a stationary assisted standing device to increase their Bone Mineral Density.
Caregiver Priorities & Child Health Index of Life with Disabilities (CPCHILD) questionnaire | 12 months
  The CPCHILD© measures caregivers' perspectives on the health status, comfort, well being, functional abilities and ease of caregiving of children with severe developmental disabilities. It was developed to measure the effectiveness of interventions intended to improve or preserve these outcomes for children with severe disabilities, including non-ambulant children with severe cerebral palsy, and traumatic or other acquired brain injuries. This will help determine if care-givers perception of health status changes with changes in standing magnitude and duration.

CONTACTS AND LOCATIONS:
Overall Officials: Walter Truong, MD, Principal Investigator — Gillette Children's Specialty Healthcare
Locations (2):
- United States (2):
  - Clinical and Translational Science Institute at University of Minnesota, Minneapolis, Minnesota
  - Gillette Children's Specialty Healthcare, Saint Paul, Minnesota